CLINICAL TRIAL: NCT00018954
Title: PILOT MULTINATIONAL PROTOCOLS IN ACUTE LYMPHOBLASTIC LEUKEMIA AND DIFFUSE NON-HODGKIN'S LYMPHOMA
Brief Title: Chemotherapy in Treating Patients With Acute Lymphoblastic Leukemia and Diffuse Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000077227; NCI-92-C-0030; NCI-T91-0259N; OH92-C-0030
Record Dates: First submitted 2001-07-11; First posted 2003-06-12 (Estimated); Last update posted 2012-02-20 (Estimated); Status verified 2012-02

CONDITIONS: Leukemia; Lymphoma
Keywords: stage I childhood lymphoblastic lymphoma; stage II childhood lymphoblastic lymphoma; stage III childhood lymphoblastic lymphoma; stage IV childhood lymphoblastic lymphoma; untreated adult acute lymphoblastic leukemia; untreated childhood acute lymphoblastic leukemia; stage I adult diffuse small cleaved cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse large cell lymphoma; stage I adult immunoblastic large cell lymphoma; stage I adult lymphoblastic lymphoma; stage I adult Burkitt lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse large cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV adult Burkitt lymphoma; stage I childhood small noncleaved cell lymphoma; stage I childhood large cell lymphoma; stage II childhood small noncleaved cell lymphoma; stage II childhood large cell lymphoma; stage III childhood small noncleaved cell lymphoma; stage III childhood large cell lymphoma; stage IV childhood small noncleaved cell lymphoma; stage IV childhood large cell lymphoma; stage I mantle cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II mantle cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult Burkitt lymphoma; contiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II mantle cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; stage I marginal zone lymphoma; stage I small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; contiguous stage II marginal zone lymphoma; contiguous stage II small lymphocytic lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Lymphoma, Non-Hodgkin; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Burkitt Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Lymphoma, Mantle-Cell; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Asparaginase; Cyclophosphamide; Cytarabine; Daunorubicin; Doxorubicin; Etoposide; Ifosfamide; Mercaptopurine; Methotrexate; Prednisone; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: asparaginase
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: doxorubicin hydrochloride
Drug: etoposide
Drug: ifosfamide
Drug: mercaptopurine
Drug: methotrexate
Drug: prednisone
Drug: vincristine sulfate
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of two treatment regimens for patients in developing countries with diffuse non-Hodgkin's lymphoma and acute lymphoblastic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Provide a standard protocol for specific therapy that is relatively easy to administer and relatively inexpensive but conforms to modern treatment principles, and determine whether such therapy can be administered safely and effectively in patients with acute lymphoblastic lymphoma or diffuse non-Hodgkin's lymphoma who live in developing countries.
* Determine the rates of relapse and survival in patients treated with these protocols, and relate this data to disease subtype and clinical presentation in order to obtain a database on which to build future stratagems.

OUTLINE: This is a multicenter study.

Patients with acute lymphoblastic leukemia or lymphoblastic lymphoma with any degree of bone marrow involvement are assigned to Protocol MCP-841. Patients with mediastinal or localized lymphoblastic lymphoma (a single nodal or extranodal site) without bone marrow involvement, or other types of diffuse non-Hodgkin's lymphoma with or without bone marrow involvement are assigned to Protocol MCP-842.

Protocol MCP-841:

* First induction therapy: Patients receive daunorubicin (DNR) IV on days 8, 15, and 29; vincristine (VCR) IV on days 1, 8, 15, 22, and 29; asparaginase (ASP) intramuscularly (IM) every other day on days 2-20; oral prednisone (PRED) on days 1-28; and methotrexate (MTX) intrathecally (IT) on days 1, 8, 15, and 22. Second induction therapy: Patients receive oral mercaptopurine (MP) on days 1-7 and 15-21; cyclophosphamide (CTX) IV over 30 minutes on days 1 and 15; MTX IT as in first induction therapy; and cranial irradiation on days 4-14.
* Alternative to second induction (if a cranial irradiation facility is unavailable): Patients receive MP and CTX as in second induction therapy; cytarabine (ARA-C) IV every 12 hours on days 1, 2, 15, 16, 29, and 30; and MTX IT on days 8 and 22.

Patients with low-risk disease (WBC no greater than 10,000/mm3, age 3 to 6 years, no prominent lymphadenopathy (less than 3 cm in diameter in each nodal region), normal CSF, no mediastinal mass, no enlargement of liver or spleen, and no cranial nerve palsies) proceed directly to maintenance therapy. All other patients are considered high risk, and they repeat first induction therapy and then proceed to consolidation therapy.

* Consolidation therapy: Patients receive MP and CTX as in second induction therapy, VCR IV on days 1 and 15, and ARA-C subcutaneously (SC) every 12 hours on days 1-3 and 15-17.
* Maintenance therapy: Patients receive VCR IV on day 1; DNR IV on day 1; oral PRED on days 1-7; ASP IM on days 1, 3, 5, and 7; and oral MTX once weekly and oral MP daily on days 15-35, 43-63, and 71-91. Maintenance therapy continues for a total of 6 courses.

Protocol MCP-842:

* Patients undergo surgical resection of intra-abdominal masses, if feasible. Patients with low-risk disease (completely resected tumor or a single extra-abdominal site of involvement (other than the mediastinum), but without lymphoblastic lymphoma) are assigned to treatment group 2. All other patients, including those with lymphoblastic lymphoma without bone marrow involvement, are considered high risk and they are assigned to treatment group 1.
* Group 1 (high risk): Patients receive one course of regimen A comprising CTX IV over 15 minutes on days 1-4; VCR IV on days 1, 8, and 15; doxorubicin (DOX) IV on days 1 and 2; ARA-C IV over 3 hours every 12 hours on day 1; ARA-C IT on day 4; and MTX IT on days 8 and 12. Patients then receive one course of regimen B comprising ifosfamide IV over 30 minutes on days 1-5, etoposide IV over 1 hour and MTX IV on days 1-3, VCR IV on day 8, ARA-C IT on days 1 and 4, and MTX IT as in regimen A. Patients then receive a second course of regimen A, followed by a second course of regimen B.
* Group 2 (low risk): Patients receive one course of regimen A, followed by one course of regimen B, and then a second course of regimen A. DOX is withheld during both courses of regimen A. IT therapy is withheld during the second course of regimen A.

Patients are followed every 2 months for 1 year (Protocol MCP-841) or at 1, 2, 3, 4, 6, and 8 months (Protocol MCP-842), every 6 months for 5 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 4,000 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed acute lymphoblastic leukemia (ALL)

  * Lymphoblasts comprising more than 25% of nucleated cells on bone marrow aspirate

    * Associated with an appropriate clinical syndrome
* OR
* Histologically proven newly diagnosed diffuse non-Hodgkin's lymphoma (NHL)
* Immunologic and/or cytochemical confirmation of diagnosis preferred

PATIENT CHARACTERISTICS:

Age:

* ALL:

  * Under 25
* NHL:

  * Not specified

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Not specified

Renal:

* Not specified

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior therapy for ALL or NHL

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1992-10; Study Completion 2002-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Trevor Magrath, MD, FRCP, FRCPath, Study Chair — National Cancer Institute (NCI)
Locations (5):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States
- National Cancer Institute of Egypt, Cairo, Egypt
- India (3):
  - Kidwai Memorial Institute of Oncology, Bangalore
  - Cancer Institute (W.I.A.), Madras
  - Tata Memorial Centre, Mumbai

REFERENCES:
- [Result] Gad-el-Mawla N, Hussein MH, Abdel-Hadi S, el-Taneer O, Adde M, Magrath I. Childhood non-Hodgkin's lymphoma in Egypt: preliminary results of treatment with a new ifosfamide-containing regimen. Cancer Chemother Pharmacol. 1989;24 Suppl 1:S20-3. doi: 10.1007/BF00253233. PMID 2758567